CLINICAL TRIAL: NCT01212731
Title: Detection of Vascular and Neuronal Changes Following Proton and/or Photon Radiotherapy in Patients Receiving Skull Base and/or Brain Radiation
Brief Title: Skull Base and Low Grade Glioma Neurocognitive Magnetic Resonance Imaging (MRI) Study
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: UPCC 08310
Record Dates: First submitted 2010-09-28; First posted 2010-10-01 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Malignancy; Glioma; Radiotherapy
Keywords: Patients with malignancies of the skull base or patients with low grade glioma who require radiotherapy.
MeSH Terms: conditions — Neoplasms; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort 1: Subjects with a histological diagnosis of malignancy of the base of skull necessitating irradiation to a minimum of 60 Gy, ECOG PS 0-1 with no evidence of metastatic disease and an estimate life expectancy of at least 1 year and who is able to provide informed consent. Subjects will undergo standard CT simulation and radiotherapy treatment planning.
  Interventions: Radiation: Photon treatment plans; Radiation: Proton Treatment Plans; Behavioral: Neurocognitive evaluation; Device: Advanced MRI imaging
- Cohort 2: Subjects with a histological diagnosis of low grade glioma requiring radiotherapy. ECOG PS 0-1 with no evidence of metastatic disease and an estimated life expectancy of at least 1 year and who is able to provide informed consent. Subjects will undergo standard CT simulation and radiotherapy treatment planning.
  Interventions: Behavioral: Neurocognitive evaluation; Device: Advanced MRI imaging

INTERVENTIONS:
Radiation: Photon treatment plans — 10 of the 30 subjects on Cohort 1 will receive photon treatment plans.
  Groups: Cohort 1
Radiation: Proton Treatment Plans — 20 subjects from Cohort 1 will receive proton treatment plans with malignancies involving the base of skull.
  Groups: Cohort 1
Behavioral: Neurocognitive evaluation — Verbal and Visual memory; immediate attention, working memory, and processing speed; executive functions and affect and depression.
Device: Advanced MRI imaging — Anatomic Imaging, Blood volume measurements, Diffusion Tensor Imaging, DTI Image Processing

SUMMARY:
The purpose of this study is to:

* estimate the degree of memory loss, if any following radiotherapy to the base of skull or brain as measured by standard neurocognitive battery testing.
* describe radiotherapy dose-related changes in vascular perfusion, in spectroscopic parameters of neuronal injury and changes in the degree and directionality of tissue water diffusivity (diffusion tensor imaging) as a measure of white axonal injury.
* to relate these imaging characteristics to the degree of memory loss.

DETAILED DESCRIPTION:
Data suggests that regions of the normal brain exposed to radiation doses that has otherwise been regarded as safe and not limited by current radiation treatment planning may contribute to the risk of late neurocognitive injury. Radiation dose-dependent subclinical vascular effects have been reported in irradiated normal brain tissue and have been hypothesized to be a potential mechanism of action. Direct neuronal injury is another potential mechanism of injury. 1)Estimate the degree of cognitive loss following RT. 2) Demonstrate evidence of radiation induced subclinical vascular and neuronal injury in adjacent brain regions receiving exit doses of radiation. Subjects will include patients with malignancies of the skull of the skull base or patients with low grade glioma who require radiotherapy. Baseline MRI imaging of the brain utilizing established techniques will be used to identify and characterize the regions of interest anatomically adjacent to the regions of intended high dose irradiation. The MRI data for the ROIs will be registered with the radiotherapy treatment planning CT in order to create a single volume of data where each voxel corresponds to a vector containing the multi-parametric information. Subsequent repeat MRI imaging will be at 1.5, 4.5, 12 and 24 months following completion of the radiotherapy for patients with low grade glioma and 1.5 and 12 months post radiotherapy for patients with malignancies involving the skull base. Both cohorts will repeat standard neurocognitive evaluation at 1.5, 4.5,12 and 24 months following completion of radiotherapy. Analysis: Neurocognitive domains will be evaluated at the designated time points.

ELIGIBILITY:
Inclusion Criteria: For Cohort 1 (Patients with tumor involving the base of skull)

* Study subjects capable of providing informed consent.
* Study subjects with an ECOG performance status of 0-1.
* Study subjects aged 18 or greater.
* Study subjects with a histological diagnosis of a malignancy of the paranasal sinuses or the nasopharynx requiring either definitive or post-operative radiation to a minimum prescribed dose of 60 Gy.
* Study subjects deemed capable of undergoing standard CT simulation and radiotherapy treatment planning and delivery including the capacity to comply with standard immobilization devices to the head and nexk for daily irradiation.
* Study subjects without any evidence of distant metastasis.
* Study subjects with an estimated life expectancy of at least 1 year.
* Study subjects who are able to receive a standard MRI study and deemed capable of complying with the immobilization needs.
* Female study subjects of reproductive potential with a negative pregnancy test prior to each scheduled MRI study.

Inclusion Criteria: For Cohort 2 (Patients with Low Grade Gliomas)

* Histological confirmed diagnosis of low grade glioma of the CNS
* WHO grade II
* Patients must have a Karnofsky Performance Status of greater than or equal to 60.
* Age greater than or equal to 18.
* Patients must be able to provide informed consent.
* Adequate bone marrow function:WBC greater than or equal to 4000/mm3, platelets greater than or equal to 100,000 mm3.
* Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms, or other barrier methods, etc.). Hysterectomy or meopause must be clinically documented.
* Study subjects deemed capable of undergoing standard CT simulation and radiotherapy treatment planning and delivery including the capacity to comply with standard immobilization devices to the brain for daily irradiation.

Exclusion Criteria: for Both Cohorts

* Study subjects with questionable performance status and in whom the treating physician is suspicious that a life expectancy of at least 1 year is possible.
* Study subjects with anxiety that precludes the safe administration of a MRI for the imaging time required.
* Study subjects with major psychiatric diagnosis prior to neuro-oncologic diagnosis.
* For neuropsychological studies, study subjects with neurological or behavioral issues that would preclude compliance with study procedures. (Karnofsky Performance Scale score of less than 60, indicating that the patients needs considerable assistance for self care and frequent medical care).
* Study subjects with an inability to undergo MR Imaging for any reason.
* Study subjects with a history of renal transplant or known renal disorder with a calculated GFR > 45mL/1min [gadolinium restriction]
* For neuropsychological studies, study subjects with mixed language background with only one year of educationin an English-speaking school.
* Pregnant women, women planning to become pregnant and women who are nursing.

Additional Exclusion Criteria for Cohort 2 (Patients with Low Grade Gliomas)

* Prior or simultaneous malignancies within the past two years (other than cutaneous squamos or basal cell carcinoma, melanoma in situ or well differentiated thyroid carcinoma).
* Patients with the following histologies are excluded: Gliomatosis cerebri, WHO III or IV gliomas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will include patients with malignancies of the skull base or patients with low grade glioma who require radiotherapy. 10 subjects receiving photon treatment plans and 20 subjects receiving proton treatment plans with malignancies involving the base skull and a total of 40 patient with low grade glioma will be prospectively enrolled.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2015-08-31 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Neurocognitive evaluation
  verbal and visual memory; immediate attention, working memory, and processing speed; executive functions and affect and depression

SECONDARY OUTCOMES:
Advance MRI imaging
  Anatomic Imaging, Blood volume measurements, Diffusion Tensor Imaging, DTI Image Processing

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Alonso Basanta, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States